CLINICAL TRIAL: NCT01528540
Title: Evaluation of Efficacy of Combination of Pregabalin and Antioxidant in Reducing Pain in Chronic Pancreatitis: a RCT
Brief Title: Evaluation of Efficacy of Combination of Pregabalin and Antioxidant in Reducing Pain in Chronic Pancreatitis: a Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIG-PAN-2012-1
Record Dates: First submitted 2012-01-27; First posted 2012-02-08 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Pancreatitis
Keywords: chronic pancreatitis; pregabalin; antioxidant
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Antioxidants; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): This group will contain a placebo for antioxidant cocktail and pregabalin
  Interventions: Drug: Placebo
- Antioxidant plus pregabalin (Experimental): This group will contain antioxidant cocktail and pregabalin
  Interventions: Drug: Antioxidant plus Pregabalin

INTERVENTIONS:
Drug: Placebo — This group will include placebo.
  Arms: Placebo
Drug: Antioxidant plus Pregabalin — This group will contain combination of antioxidant cocktail and pregabalin
  Arms: Antioxidant plus pregabalin

SUMMARY:
Study hypothesis: Combination of antioxidants and pregabalin results in better pain relief than placebo in patients with chronic pancreatitis.

Chronic pancreatitis (CP) is a clinical enigma, with pain being the most distressing symptom that brings the patient to clinical attention. Pain in chronic pancreatitis is multifactorial, and may be related to pancreatic ductal hypertension, tissue hypertension, inflammatory cytokines, oxidative stress and neuropathic mechanisms like mechanical allodynia, inflammatory hyperalgesia and temporal summation. The mainstay of treatment for pain in CP due to pancreatic ductal stone is endotherapy (ESWL and ERCP). Recent randomized controlled trials have shown that antioxidant cocktail and pregabalin (a presynaptic voltage gated calcium channel blocking agent) can result in significant reduction of pain in CP.

In this study, the investigators will study the efficacy of the combination of antioxidants and pregabalin in reducing pain and compare that with placebo. The investigators will randomize patients with documented chronic pancreatitis with recurrent/persistent pain after undergoing endotherapy and ductal clearance into three groups: Group A- antioxidants + pregabalin; Group B- Placebo. The primary outcome will be change in pain score and the secondary outcomes will be change in the number of painful days, analgesic requirements, quality of life and depression scale. Pain score will be quantified by the Izbicki pain score and visual analog scale; while quality of life and depression will be measured by the EORTC QLQ-C30/PAN26 and Beck depression inventory respectively. Comparison between Group A vs B will be made by the Chi square test/Fischer Exact and the Student's 't' tests respectively and analysis will be done on a intention to treat and per protocol basis. With an expected improvement of pain by 40% (at 80% power and alpha of 0.05) and adjusting for a presumed 10% drop out rate, the required sample size in each group will be at least 40.

ELIGIBILITY:
Inclusion Criteria:

1. Epigastric pain +/- radiation at least thrice in one month over the past three month.
2. Endotherapy/Surgery and ducal clearance

Exclusion Criteria:

1. Age <18 and >65yrs
2. MPD and biliary obstruction
3. Pancreatic neoplastic lesions
4. Acute flare
5. Pancreatic pseudocysts
6. Pregnancy
7. Cardiac and renal diseases
8. Use of other anti epileptics
9. Hypersensitivity to gabapentin/pregabalin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in the pain score | Baseline and 8weeks
  Pain score will be assessed by the Izbicki pain score, Visual analog scale and painDETECT tool for neuropathic pain.

SECONDARY OUTCOMES:
Change in number of painful days | Baseline and 8weeks
  The number of days of pain per week will be measured.
Change in analgesic requirement | Baseline and 8weeks
  The type (opiate/non-opiate), number and route of additional analgesic medicines that were required within the study period will be evaluated.
Change in quality of life | Baseline and 8weeks
  QOL will be evaluated with the EORTC QLQ-C30/PAN26 questionnaire
Change in depression scale | Baseline and 8weeks
  Depression will be assessed with the Beck's Depression Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Rupjyoti Talukdar, MD, Principal Investigator — Asian Institue of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Andhra Pradesh, India

REFERENCES:
- [Background] Bhardwaj P, Garg PK, Maulik SK, Saraya A, Tandon RK, Acharya SK. A randomized controlled trial of antioxidant supplementation for pain relief in patients with chronic pancreatitis. Gastroenterology. 2009 Jan;136(1):149-159.e2. doi: 10.1053/j.gastro.2008.09.028. Epub 2008 Sep 25. PMID 18952082
- [Background] Olesen SS, Bouwense SA, Wilder-Smith OH, van Goor H, Drewes AM. Pregabalin reduces pain in patients with chronic pancreatitis in a randomized, controlled trial. Gastroenterology. 2011 Aug;141(2):536-43. doi: 10.1053/j.gastro.2011.04.003. Epub 2011 Apr 14. PMID 21683078